CLINICAL TRIAL: NCT02481492
Title: Randomized Controlled Trial of Shang Ring Male Children Circumcision: Comparison Between Flip and No Flip Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Collaborators: The Affiliated Hospital of Medical College, Ningbo University (Other)
Responsible Party: Principal Investigator, Li Fang, M.D., Ningbo No. 1 Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: NBDYYY2015001
Record Dates: First submitted 2015-06-22; First posted 2015-06-25 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Human Immunodeficiency Virus
Keywords: Circumcision, Male; Shang Ring; Children; Foreskin
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No flip technique (Experimental): One group of boys will undergo a circumcision with no flip technique of Shang Ring Circumcision and receive regular follow-up to evaluate pain, operation associated adverse events, wound healing time. The Shang Ring will detach spontaneously without intervention, and the participants are asked to have a visit soon after ring detached. The last scheduled follow-up visit is at 90 days.
  Interventions: Device: No flip technique of Shang Ring circumcision
- Flip technique (Experimental): One group of boys will undergo a circumcision with flip technique of Shang Ring Circumcision and receive regular follow-up to evaluate pain, operation associated adverse events, wound healing time. The Shang Ring will be removed at 7 days, and the last scheduled follow-up visit is at 90 days.
  Interventions: Device: Flip technique of Shang Ring circumcision

INTERVENTIONS:
Device: No flip technique of Shang Ring circumcision — Measure the diameter of the penis with a scale plate of holes, the diameter of the ring was accordance with the glands, inner ring is placed into foreskin cavity, apply the outer ring on the skin covering inner ring, clamp the out ring and cut the redundant foreskin; Ring is detached spontaneously.
  Arms: No flip technique
Device: Flip technique of Shang Ring circumcision — Measure the diameter of the penis with a scale plate of holes, the diameter of the ring was accordance with the penis, inner ring is placed around the penis, flip foreskin over the inner ring, apply the outer ring on the skin covering inner ring, clamp the out ring and cut the redundant foreskin; Remove the ring 7days postoperatively.
  Arms: Flip technique

SUMMARY:
This is a prospect, randomized control trial to evaluate merits between flip and no flip technique in Shang Ring children circumcision.

DETAILED DESCRIPTION:
The boys between 7 and 12 years old seeking for circumcision in The Affiliated Hospital of Medicine School of Ningbo University will be evaluated. Those who match the inclusion criteria and without exclusion criteria will be recruited.

The investigators will perform randomization preoperatively. participants were distributed into No Flip Group and Flip Group correspondingly according to a table of random number.

All of the procedures will be performed by a specific study surgeon in the hospital operation room. An assistant will take the pictures and recorder the parameters needed. In both groups, participants will be measured twice by a scale plate of holes, the diameter of penis with the foreskin noneverted and the diameter of exposed glans. Local anesthesia will be administered to the dorsal penile nerve using 2% lidocaine. The operation will not begin until the anesthesia is satisfied. The proper ring will be chosen according to different strategies of two groups. Participants will stay in hospital for 24 hours after operation. Pain during operation, half a hour post-operation and 24 hours will be evaluated, adverse events at hospital will be recorded carefully as well.

Participants will be advised to return usually at 7th, 14th, 21st, 28th and 90th post-operative days. However, if the wound does not heal completely 28 days post-operatively, the participant will be asked come to visit weekly until complete healing. All of the assessments will be performed and recorded by the lead investigator.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 7 years and 12 years(inclusive);
* Must be accompanied by the parent or legally acceptable representative (LAR), who freely agrees with participation of the child into the study;
* Must tolerate local anesthesia;
* Must be in good general health;
* Parent or LAR and if possible the client must be able to understand study procedures and requirements of study participation;
* Parent or LAR must agree to return the client to the study site for the full schedule of follow-up visits after his circumcision;
* Parent or LAR must agree the study staff to take photos during operation or follow-up if necessary, and
* Parent or LAR must agree to provide the study staff with an address, phone number, or other locator information

Exclusion Criteria:

* Has a known allergy or sensitivity to lidocaine or other local anesthesia;
* Takes a medication that would be a contraindication for elective surgery (e.g anticoagulant , steroid);
* Has known bleeding/clotting disorder (e.g. hemophilia);
* Has an active genital infection, anatomic abnormality or other condition(e.g. concealed penis, hypospadias, epispadia, micropenis);
* Is currently participating in another biomedical research study; or
* Participants under other condition (e.g. severe obesity, diabetes or sickle cell anemia) should be excluded from this study in the opinion of the surgeon.

Ages: 7 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain score on the Visual Analog Scale | 28 days
  The pain during and after the two circumcision methods will be compared. Visual Analogue Scale(VAS) will be used to evaluate the pain during operation, 30min post-operatively, 24h post-operatively, ring detachment and during the recovery period.
Adverse events | 3 months
  The adverse events such as edema, wound infection, bleeding, unsymmetrical foreskin, wound dehiscence will be recorded.

SECONDARY OUTCOMES:
Time to complete healing | 3 months
  The healing time will be observe by study primary investigator. The usually following time is once a week during the first month and then 3 months later. However, if the wound does not heal completely 28 days post-operatively, the participant will be asked come to visit weekly until complete healing.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Cheng, MD, Principal Investigator — Ningbo No. 1 Hospital; Jianhua He, MD, Study Director — The Affiliated Hospital of Medical College, Ningbo University
Locations (2):
- China (2):
  - The Affiliated Hospital of Medical College, Ningbo University, Ningbo, Zhejiang
  - Ningbo NO.1 hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yue C, Ze-Jun Y, Wu KR, Su XJ, Hu JS, Ma JW, Guo CM, Fang HW, Su R, Zhang Y, Zhang QH. A randomized clinical study of circumcision with a ring device versus conventional circumcision. J Urol. 2012 Nov;188(5):1849-54. doi: 10.1016/j.juro.2012.07.048. Epub 2012 Sep 19. PMID 22999700 (Retraction: PMID 23293788 J Urol. 2012 Dec;188(6):2443)
- [Background] Cheng Y, Peng YF, Liu YD, Tian L, Lu NQ, Su XJ, Yan ZJ, Hu JS, Lee R, Kim HH, Sokal DC, Li PS. [A recommendable standard protocol of adult male circumcision with the Chinese Shang Ring: outcomes of 328 cases in China]. Zhonghua Nan Ke Xue. 2009 Jul;15(7):584-92. Chinese. PMID 19694369
- [Background] Yan B, You H, Zhang K, Tang HY, Mao W, He GH, Yin ZG. [Circumcision with the Chinese Shang Ring in children: outcomes of 824 cases]. Zhonghua Nan Ke Xue. 2010 Mar;16(3):250-3. Chinese. PMID 20369555
- [Background] Barone MA, Awori QD, Li PS, Simba RO, Weaver MA, Okech JO, Aduda AO, Cherutich P, Muraguri N, Wekesa JM, Nyanchoka J, Perchal P, Masson P, Lee R, Goldstein M, Kioko J, Lusi O, Sokal DC. Randomized trial of the Shang Ring for adult male circumcision with removal at one to three weeks: delayed removal leads to detachment. J Acquir Immune Defic Syndr. 2012 Jul 1;60(3):e82-9. doi: 10.1097/QAI.0b013e31824ea1f2. PMID 22343180
- [Background] Masson P, Li PS, Barone MA, Goldstein M. The ShangRing device for simplified adult circumcision. Nat Rev Urol. 2010 Nov;7(11):638-42. doi: 10.1038/nrurol.2010.167. Epub 2010 Oct 12. PMID 20938437
- [Background] Cheng Y, Wu K, Yan Z, Yang S, Li F, Su X. Long-term follow-up for Shang Ring male circumcision. Chin Med J (Engl). 2014;127(10):1879-83. PMID 24824249
- [Background] Cheng Y, Wu K, Yan Z, Guo C, Ma J, Su X, Yang S. How to choose appropriate ring size for Shang Ring male circumcision. J Acquir Immune Defic Syndr. 2012 Dec 15;61(5):606-9. doi: 10.1097/QAI.0b013e318273aec9. PMID 23018373
- [Background] Pan L, Zhang A, Shen R, Wang Z. Acceptability of early infant male circumcision among Chinese parents: strategy implications of HIV prevention for China. BMC Public Health. 2012 Sep 4;12:738. doi: 10.1186/1471-2458-12-738. PMID 22946988
- [Background] Peng YF, Cheng Y, Wang GY, Wang SQ, Jia C, Yang BH, Zhu R, Jian SC, Li QW, Geng DW. Clinical application of a new device for minimally invasive circumcision. Asian J Androl. 2008 May;10(3):447-54. doi: 10.1111/j.1745-7262.2008.00411.x. PMID 18385906
- [Background] Wu X, Wang Y, Zheng J, Shen W, Yan JA, Ji H, Li X, Zhang H, Zhou Z. A report of 918 cases of circumcision with the Shang Ring: comparison between children and adults. Urology. 2013 May;81(5):1058-63. doi: 10.1016/j.urology.2012.11.046. Epub 2013 Mar 7. PMID 23465168